CLINICAL TRIAL: NCT02663219
Title: Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected Men Who Have Sex With Men (MSM) in the United States
Brief Title: Enhancing Recruitment, Linkage to Care and Treatment for HIV-Infected MSM in the United States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 078; UM1AI068619 (NIH); 11995 (Other: DAIDS)
Record Dates: First submitted 2016-01-13; First posted 2016-01-26 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: HIV
Keywords: MSM; ART; CCM; DAIDS; HPTN; ACA; PAF; PEP; RDS
MeSH Terms: interventions — Methods; Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will provide a Case Manager (CM) intervention package designed to enhance linkage to care, antiretroviral treatment (ART) initiation, treatment adherence and retention in care.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Intervention — The intervention arm will provide a Case Manager (CM) intervention package designed to enhance linkage to care, antiretroviral treatment (ART) initiation, treatment adherence and retention in care.
  Other Names: Case Management
  Arms: Intervention

SUMMARY:
The purpose of this study is to develop and assess the efficacy of an integrated strategy that includes feasible and scalable interventions to identify, recruit, link to care, retain in care, attain, and maintain viral suppression among HIV-infected men who have sex with men (MSM) in the United States (US).

DETAILED DESCRIPTION:
This study will use deep-chain respondent driven sampling (DC-RDS) and direct recruitment (DR) to identify and recruit HIV-infected MSM who are not virally suppressed. A subset of these men will be enrolled into one of two study arms. The intervention arm will provide a Case Manager (CM) intervention package designed to enhance linkage to care, antiretroviral treatment (ART) initiation, treatment adherence and retention in care. The control arm will provide the standard of care (SOC) for linkage to care, initiation of ART, treatment adherence and retention in care. The primary outcome of the study is viral suppression 12 months after enrollment. Phylogenetic methods will be used to evaluate the relationship between viruses in study participants. Mathematical modeling will be performed using demographic, behavioral, and clinical data generated from this study and other sources to estimate the population-level impact of the CM intervention on HIV incidence and to estimate the level of identification, linkage, ART coverage and viral suppression that would be required to achieve a substantial reduction in HIV incidence among MSM in the US settings where the study is conducted.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for study screening:

* Biological male (at birth)
* Self-report of history of anal intercourse with another man
* 16 years or older

Individuals who are eligible for screening and who meet all of the following criteria are eligible for enrollment into the CM intervention and SOC control arms:

* HIV-infected, as defined in the HPTN 078 Study-Specific Procedures (SSP) Manual
* Not virally suppressed (defined as HIV VL ≥ 1000 copies/ml)
* Can receive HIV care at one of the participating clinics (as chosen by each site)
* No current plan to relocate in the 24 months following enrollment

Exclusion Criteria:

Individuals who meet any of the following criteria will be excluded from study screening:

* Unable or unwilling to provide consent/assent for study participation.
* Active or previous participation in an HIV vaccine trial.
* Any condition that, in the opinion of the Investigator of Record (IoR), would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Individuals who are eligible for screening, but who meet the following criteria are excluded from enrollment into the CM intervention and SOC control arms:

• Current participation in a linkage or ART adherence study

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — biologically male
Enrollment: 144 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
HIV status at screening for each MSM recruited | At Baseline
  HIV status
HIV viral load at screening for each MSM recruited | 12 months
  HIV viral load
HIV viral load at month 24 of participants randomized | 24 months
  time driven HIV viral load

SECONDARY OUTCOMES:
Date of recruitment for each man recruited by DC-RDS | During recruitment period
  recruitment timeline
Wave of recruitment for each man recruited by DC-RDS | During recruitment period
  recruitment timeline
HIV viral load of those randomized | HIV viral load at Months 3, 6, 9, 12
  HIV viral load
Number of all care visits from randomization through the end of 12 months follow up | Over 12 months
  clinical care uptake
Time of all care visits from randomization through the end of 12 months follow up | Over 12 months
  clinical care uptake
HCV status at baseline | At Baseline
  HCV status
Baseline Demographics | At Baseline
  Participant-administered questionnaire
CD4 status at baseline | At Baseline
  CD4 cell count
HIV viral load status at baseline | At Baseline
  HIV viral load
Syphilis status at baseline | At Baseline
  Syphilis status
Self-reported sexual risk behavior of unprotected anal intercourse, characteristics of 3 most recent partners) at baseline and 24 months | 12 months
  participant-administered questionnaire

OTHER OUTCOMES:
Health care utilization at baseline and 24 months | Up to 24 months
  computer assisted self interview
Stigma at baseline and 24 months | Up to 24 months
  computer assisted self interview
Number of contacts (text message, email, phone, in person) for each participant randomized to the CM intervention arm over follow-up | Up to 24 months
  clinical contact
Open-ended questions for process evaluation | Up to 12 months
  Open ended qualitative data compiled and coded
The phylogenetic relationship between HIV sequences | Up to 24 months
  HIV genetic sequencing
Syphilis positive or negative at baseline | Up to 24 months
  STI description at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chris Beyrer, MD/MPH, Study Chair — Johns Hopkins University; Robert H Remien, PhD, Study Chair — Columbia University
Locations (4):
- United States (4):
  - Alabama CRS, Birmingham, Alabama
  - Ponce de Leon CRS, Atlanta, Georgia
  - Johns Hopkins Baltimore CRS, Baltimore, Maryland
  - Fenway Health CRS, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] KM Mitchell, B Hoots, D Dimitrov, et al. Potential Impact on HIV Incidence of Increasing Viral Suppression among HIV- positive MSM in Baltimore: Mathematical Modelling for HPTN 078. HIV Research for Prevention (HIVR4P 2016). Chicago, October 17-21, 2016. Abstract OA10.04
- [Derived] Maragh-Bass AC, Hucks-Ortiz C, Beyrer C, Remien RH, Mayer K, Del Rio C, Batey DS, Farley JE, Gamble T, Tolley EE. Multilevel Stigma and Its Associations with Medical Care Ratings Among Men Who Have Sex With Men in HPTN 078. J Prim Care Community Health. 2023 Jan-Dec;14:21501319231175362. doi: 10.1177/21501319231175362. PMID 37243342
- See also: Potential Impact on HIV Incidence of Increasing Viral Suppression among HIV- positive MSM in Baltimore: Mathematical Modelling for HPTN 078 — https://www.hptn.org/sites/default/files/2016-10/R4P_slides_KM_078_modelling_181016_FINAL.pdf

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT02663219/Prot_ICF_000.pdf